CLINICAL TRIAL: NCT07005271
Title: Investigation of the Effects of Virtual Reality-Based Hand Exercises on Cognitive Function and Hand Dexterity in Older Adults With Mild Cognitive Impairment.
Brief Title: VR Hand Exercises: Impact on Cognition and Dexterity in MCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-326
Record Dates: First submitted 2025-06-03; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: virtual reality; hand exercise; mild cognitive impairment; cortical activation; hand dextery
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (Experimental): Participants in this group will perform hand exercises using virtual reality. They will complete task-oriented hand exercises resembling activities of daily living through the ErgoActive system, which consists of four different games.
  Interventions: Behavioral: virtual reality
- Conventional treatment (Active Comparator): Participants in this group will perform exercises involving hand skills used in daily life. These exercises will be similar to those in the virtual reality group but will be carried out in their real-life form.
  Interventions: Behavioral: Conventional treatment

INTERVENTIONS:
Behavioral: virtual reality — The exercises in this group consist of four different games, including: (1) MasterChef, which involves performing daily living tasks in a virtual kitchen environment such as slicing tomatoes and cheese, adding salt, cracking and adding eggs, and stirring with a fork to prepare an omelet; (2) PinchPeg, where participants use a pinch grip to grasp rods generated in the center of a virtual environment and place them into holes on a pegboard, followed by removing and returning them to their original location; (3) Hold and Put, which requires the use of a standard palmar grasp to pick up virtual cups or cans and place them onto designated shelves; and (4) bPuzzle, a task that integrates cognitive and fine motor exercises by requiring participants to change the color of a puzzle using finger movements and place the pieces into the correct positions using hand gestures.
  Arms: virtual reality
Behavioral: Conventional treatment — Participants will be asked to complete puzzles consisting of 30 to 50 pieces, with 3 to 4 different puzzles used to eliminate the learning effect. They will perform the Nine-Hole Peg Test, which is similar to the PinchPeg game in the virtual reality group, by picking up pegs one by one from a container and placing them into holes on the board as quickly as possible using only the evaluated hand; this will be used for training purposes. Additionally, participants will be instructed to cut out geometric shapes with dotted outlines using scissors, aiming to follow the lines accurately. Finally, they will sort objects by placing the correct number and color of items into designated locations according to a predetermined pattern, and use a magnetic fishing rod to catch wooden fish, promoting both fine motor skills and task-oriented hand function.
  Arms: Conventional treatment

SUMMARY:
This study aims to investigate the effects of virtual reality (VR)-based hand exercises on cognitive functions and hand skills in older adults with mild cognitive impairment (MCI). Cognitive functions will be assessed by measuring brain activity using functional near-infrared spectroscopy (fNIRS) during the Stroop test. Additionally, hand functions will be evaluated using the Minnesota Manual Dexterity Test, grip strength measurement (via a Jamar dynamometer), and the Duruöz Hand Index. Hand dominance will be determined using the Edinburgh Handedness Inventory, and sociodemographic data will be collected through a form prepared by the researcher. Based on a G*Power analysis, a total of 30 participants-15 in each group-will be included in the study, with an effect size of 1.00094 and a power of 80%. Evaluations will be conducted twice, before and after the intervention. To avoid participant fatigue, assessments will be divided over two days. The intervention group will receive VR-based hand exercises twice a week for six weeks. These exercises will include activities such as MasterChef (cutting, mixing, and grasping in a virtual kitchen), PinchPeg (placing pegs using pinch grip), HoldAndPut (transporting cups or cans), and bPuzzle (color matching and puzzle completion). The control group will perform traditional exercises twice a week for six weeks, including 30-50 piece puzzle completion, the Nine-Hole Peg Test, shape cutting, and number-color matching tasks. The study will be conducted with volunteer participants at the Istanbul Metropolitan Municipality Darülaceze Directorate, and written and verbal informed consent will be obtained from all participants in accordance with the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 65 and 75 years.
* Diagnosed with mild cognitive impairment by the institution's physician during routine examination.
* Ability to understand and follow verbal instructions.

Exclusion Criteria:

* Presence of neurodegenerative diseases affecting cognitive functions.
* Auditory or visual impairments that could interfere with rehabilitation implementation and communication.
* Upper extremity disorders, including severe shoulder, elbow, wrist, or finger impairments, bilateral elbow, hand or wrist fractures, or advanced rheumatoid arthritis.
* Participation in any rehabilitation program during the study period.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Cortical Hemodynamics (Functional Near-Infrared Spectroscopy) | before treatment, week 6
Hand skills (Minnesota Manual Dexterity Test) | before treatment, week 6
Activities of daily living (Duruöz Hand Index) | before treatment, week 6

SECONDARY OUTCOMES:
Gross grip strength (Jamar hand dynamometer) | before treatment, week 6
Determination of hand preference (Edinburgh Handedness Inventory) | before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Berrak Varhan, Study Chair — Istinye University

IPD SHARING:
Plan to Share IPD: Yes
The study will share de-identified, summary-level outcome data, including group-level means, standard deviations, effect sizes, and p-values derived from statistical analyses. These data will be provided to support transparency and allow for interpretation of the study findings.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Summary-level data and supporting documents (e.g., study protocol and statistical analysis plan) will be available within 12 months following the final publication of study results and will remain accessible for at least 5 years via institutional repository or upon reasonable request.
Access Criteria: The study's outcome results, including group-level means, standard deviations, p-values, and effect sizes, as well as supporting materials such as the study protocol and statistical analysis plan, will be made available to qualified academic researchers upon reasonable request. Data will be provided for ethically approved, non-commercial research purposes. Interested investigators should contact the principal investigator through the affiliated institution and submit a written request describing the intended use and data handling procedures. Each request will be reviewed individually in accordance with institutional data-sharing guideline.

REFERENCES:
- [Background] Park JH. Effects of Cognitive-Physical Dual-Task Training on Executive Function and Activity in the Prefrontal Cortex of Older Adults with Mild Cognitive Impairment. Brain Neurorehabil. 2021 Sep 13;14(3):e23. doi: 10.12786/bn.2021.14.e23. eCollection 2021 Nov. PMID 36741221
- [Background] Liao YY, Tseng HY, Lin YJ, Wang CJ, Hsu WC. Using virtual reality-based training to improve cognitive function, instrumental activities of daily living and neural efficiency in older adults with mild cognitive impairment. Eur J Phys Rehabil Med. 2020 Feb;56(1):47-57. doi: 10.23736/S1973-9087.19.05899-4. Epub 2019 Oct 15. PMID 31615196